CLINICAL TRIAL: NCT04545918
Title: Assessing a Mask Region-based Convolutional Neural Network in Follicle Identification and Measurement During Ovarian Stimulation
Brief Title: Convolutional Neural Network in Ovarian Follicle Identification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cycle Clarity (Industry)
Responsible Party: Sponsor
Other Study IDs: CC2020-001
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Infertility, Female; Ovarian Follicular Cyst
Keywords: Infertility; Ovarian Follicle
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Infertile Female: 90 female patients with infertility undergoing an ovarian stimulation with use of exogenous gonadotropins.
  Interventions: Device: Follicle Clarity

INTERVENTIONS:
Device: Follicle Clarity — Mask Region-based Convolutional Neural Network in Ultrasound Follicle Identification

SUMMARY:
A prospective cohort trial studying patients with infertility undergoing an ovarian stimulation with exogenous gonadotropins. Ovarian monitoring will be performed with a combination of transvaginal ultrasound and 2 dimensional human measurements of the follicle development on the right and left ovaries along with SonoAVC. Human and SonoAVC measurements will then be compared to mask region-based convolutional neural network in follicle identification and measurement during during the ovarian stimulation.

DETAILED DESCRIPTION:
This is a prospective cohort trial in which a total of 80 female subjects with infertility between the ages of 21 and 42 years of age undergoing ovarian stimulation will be recruited. After giving informed written consent the subject to undergo standard ovarian ultrasound monitoring with transvaginal ultrasounds during the ovarian stimulation. Monitoring will be performed with two-dimensional measurements of each follicle greater than 10 mm in size by the ultrasonographer. SonoAVC will then be applied to both ovaries for automated counting and measurement of the follicles within the ovaries. The patient will then undergo two 6-second ultrasounds of the right and left ovaries which will then be transmitted in a DICOM format to mask regional based recurrent neural network which is been trained and validated for follicle detection and quantification using curated transvaginal ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women ages 21-42 years old undergoing ovarian hyperstimulation as part of the treatment care.

Women with at least one ovary visible with transvaginal ultrasound. Women with at least one follicle 10 mm or greater in average diameter.

Exclusion Criteria:

* Women less than 21 years of age or greater than 42 years of age. Women without a visible ovary by transvaginal ultrasound. Women without a follicle at least 10 mm in average diameter

Ages: 21 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Eighty (80) consecutive female subjects of any race, 21 - 42 years of age meeting the inclusion criteria will be enrolled in the study conducted at one of 4 Coastal Fertility Specialists fertility clinics located in South Carolina and Georgia, USA.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Median size (mm) of ovarian follicles in CCAI compared to SonoAVC | 1 month
  Comparison of the mean size in mm of Cycle Clarity's Artificial Intelligence software (CCAI) compared with GE SonoAVC

SECONDARY OUTCOMES:
Number of ovarian follicles in CCAI compared to Sono | 1 month
  Comparison of the number of ovarian follicles with Cycle Clarity's Artificial Intelligence software (CCAI) compared with GE SonoAVC

CONTACTS AND LOCATIONS:
Overall Officials: John A. Schnorr, MD, Study Chair — Cycle Clarity, Founder
Locations (1):
- Coastal Fertility Specialists, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Inany HG, Youssef MA, Ayeleke RO, Brown J, Lam WS, Broekmans FJ. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD001750. doi: 10.1002/14651858.CD001750.pub4. PMID 27126581
- [Background] Gordon K, Hodgen GD. GnRH analogues in ovarian stimulation. Ann N Y Acad Sci. 1991;626:238-49. doi: 10.1111/j.1749-6632.1991.tb37919.x. No abstract available. PMID 2058957